CLINICAL TRIAL: NCT02602873
Title: Guangzhou Women and Children's Medical Center
Brief Title: Study of Tacrolimus Used for Pediatric Patients With Nephrotic Syndrome Based on Pharmacogenomics and Metabonomics
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Mo Xiaolan, Clinical Pharmacist, Guangzhou Women and Children's Medical Center
Other Study IDs: 683292136
Record Dates: First submitted 2015-09-09; First posted 2015-11-11 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — DNAs extracted from whole blood are stored in freezer with -80 centigrade.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- good efficacy: using therapeutic drug monitoring to adjust the dose of tacrolimus. patients can reach effective outcome.
  Interventions: Other: therapeutic drug monitoring
- poor efficacy: using therapeutic drug monitoring to adjust the dose of tacrolimus. patients can not reach effective outcome.
  Interventions: Other: therapeutic drug monitoring

INTERVENTIONS:
Other: therapeutic drug monitoring — with therapeutic drug monitoring , dose of tacrolimus can be adjusted by therapeutic drug monitoring.

SUMMARY:
Tacrolimus is recommended to be the first line therapeutic medication within the several immunosuppressive agents when treating refractory pediatric nephrotic syndrome, because of its definite efficacy and low toxicity. But there are still some key problems which hinder the using of tacrolimus in clinic, such as its narrow therapeutic widow, great individual difference of pharmacokinetics. Routine therapeutic drug monitoring(TDM) is needed in practice. But the disadvantage of TDM is hysteresis, which could lead to treatment failure or toxicity. To find out the reasons of great pharmacokinetic difference between patients and find out the individual proper dosage before administration are important for the clinical using of tacrolimus.

It is hot in research of tacrolimus in organ transplant field, such as the association between gene polymorphisms of cytochrome P-450 3A4, 3A5 and multiple drug resistant gene(MDR1) and concentration of tacrolimus. However, there is few study about pharmacogenomics and metabonomics of tacrolimus in patients of nephrotic syndrome.

The aim is to study the relationships between pharmacogenomics, metabonomics of tacrolimus and its efficacy, toxicity and blood concentration in patients of nephrotic syndrome, to find out the exact dosage before administration, to provide reference to individual drug administration.

DETAILED DESCRIPTION:
Investigators will collect data about efficacy and adverse drug reaction(ADR) such as time of efficacy when evaluated, how to evaluate ADR, data of demography, etc.

ELIGIBILITY:
Inclusion Criteria:

1. patients with refractory nephrotic syndrome;
2. patients age ≤14y.

Exclusion Criteria:

1. patients are sensitive to steroid;
2. combined therapy with other immunosuppressive agent;
3. combined using drugs which maybe interact the concentration of tacrolimus;
4. with other malignant disease, such as tumor.

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients with nephrotic syndrome
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
"Genotypes as measured by polymerase chain reaction-restriction fragment length polymorphism" | 1 week
  genotype are collected from hospital system.
"Concentration as measured by liquid chromatography mass spectrometry" | 1 week
  concentration of tacrolimus are collected from hospital system.
"Relationship between genotypes and concentration as analyzed at 1 week" | 1 week
  using Statistic Package for Social Science 21.0 software to analyze the relationship between gene polymorphism and concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Min Huang, Doctor, Study Director — Sun Yat-sen University
Locations (1):
- Guangzhou women and children's medical center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
we are carrying out experiment now. Data is not ready to publish for not completing the study. We will share data when we complete our study.

REFERENCES:
- [Derived] Mo X, Li J, Liu Y, Liao X, Tan M, Chen Y, He F, He Y, Li Y, Huang M. Kidney podocyte-associated gene polymorphisms affect tacrolimus concentration in pediatric patients with refractory nephrotic syndrome. Pharmacogenomics J. 2020 Aug;20(4):543-552. doi: 10.1038/s41397-019-0141-x. Epub 2020 Jan 6. PMID 31902946